CLINICAL TRIAL: NCT06264089
Title: Effects of Preservation Rhinoplasty Nasal Valve Angle and Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yaser Said Cetin, Associate Professor, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202015
Record Dates: First submitted 2023-09-28; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Nasal Obstruction, Bilateral
MeSH Terms: conditions — Nasal Obstruction | interventions — Amino Acid Motifs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No Arms have been specified for this study (Other): No Arms have been specified for this study
  Interventions: Procedure: Preservation Rhinoplasty Nasal Valve Angle and Area

INTERVENTIONS:
Procedure: Preservation Rhinoplasty Nasal Valve Angle and Area — The same group of patients who underwent Preservation Rhinoplasty will be followed and the nasal valve angles before and after surgery will be compared.
  Other Names: Preservation Rhinoplasty

SUMMARY:
The study planned to compare the internal nasal valve angle measurements of patients who underwent preservation rhinoplasty before and after surgery.

DETAILED DESCRIPTION:
Nasal congestion is one of the most common complaints in Otorhinolaryngology medicine. One of the most common causes of this is the collapse or blockage of the Internal Nasal Valve (INV). The internal nasal valve is the narrowest part of the airway and creates the greatest resistance to airflow. Its most important function is to regulate the inspiratory airflow. It is determined by the angle formed between the caudal part of the upper lateral cartilage and the nasal septal cartilage. This angle normally varies between 9-15 degrees. The tip of the inferior turbinate and the tissues surrounding the piriform aperture may affect this area. When this angle is less than 9 degrees, the valve collapses in inspiration. The internal nasal valve region should be evaluated in every patient complaining of nasal congestion. the investigators planned to radiologically examine the improvement in the internal nasal valve angle of the patients we operated on.

ELIGIBILITY:
Inclusion Criteria:

* Preservation rhinoseptoplasty

Exclusion Criteria:

* Absence of nasal obstruction
* Previous nasosinusal surgery
* Cranio-facial anomalies
* Presence of nasosinusal tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation Scale (NOSE) | 12 month
  Nasal Obstruction Symptom Evaluation Scale (NOSE)
  The NOSE will be used to measure the quality of life related to nasal obstruction. It is a validated instrument specifically designed for use in patients with nasal obstruction. According to this scale patients are asked to evaluate difficulty breathing in a general way and specifically the difficulty in breathing through the nose, breathing during sleep, and severity of their nasal congestion. The severity of the symptoms is recorded on a scale of 0 to 4, with 0 being the absence of a problem and 4 being a serious problem. The possible scores range from 0 to 20 and the higher scores indicate a higher degree of nasal obstruction. The sum of the scores is multiplied by 5 so as to obtain a final score ranging from 0 to 100, with higher values associated with poorer quality of life. The scale will be applied at the base line and at the end of 12 months.

SECONDARY OUTCOMES:
Reformatted coronal Computed tomography | 12 month
  The internal and external nasal valve levels of patients scheduled for septorhinoplasty surgery will be prospectively examined preoperatively and postoperatively with a high-resolution 3-plan (axial-sagittal-coronal) CT study. Axial CT studies will be obtained with the latest generation, 128-channel, multi-slice CT scanners (Siemens SOMATOM Definition AS+128, Forchheim, Germany) with a slice thickness of 0.5 to 1.25 mm in the bone algorithm. Axial slices will be acquired from the top of the frontal sinuses to the bottom of the maxillary incisors. Studies will be made from random selections and without correlation to diagnosis or indication.
  Axial data will be transferred to the workstation (Siemens Syngo Via Workstation) for postprocessing and measurements will be performed on this workstation.

CONTACTS AND LOCATIONS:
Locations (1):
- Yaser Said Cetin, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No